CLINICAL TRIAL: NCT05659862
Title: Efficacy of Digitally Assisted Behavioral Physical Activity Intervention in Fibromyalgia Syndrome
Brief Title: Digitally Assisted Behavioral Physical Activity Intervention in Fibromyalgia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Nimet Sermenli, Research Assistant, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09.2022.603
Record Dates: First submitted 2022-12-01; First posted 2022-12-21 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Fibromyalgia; Physical Inactivity
Keywords: fibromyalgia; physical activity; digital health; physical activity intervention
MeSH Terms: conditions — Fibromyalgia; Sedentary Behavior; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digitally assisted behavioral physical activity intervention+Education (Experimental): An activity diary and a pedometer will be given to write down the number of steps per day.
  After one week, the patient will be asked to send the activity diary as a photo via WhatsApp.
  Afterwards, a 20-minute phone call will be made to provide patient education.
  After the patient education, the patient will be consulted about the average number of steps he wants to take at the end of the intervention, and the daily average number of steps will be determined for the first week of the intervention, taking into account the patient's number of steps in the last week and the goal of the number of steps she wants to reach.
  The person will be added to the WhatsApp patient support group. Patients will receive messages from this group by the researcher twice a week.
  The target for the number of steps will be renewed every next week and an average of 20 minutes of phone calls including motivational interviews will be held in the light of Social Cognitive Theory.
  Interventions: Behavioral: Digitally assisted behavioral physical activity intervention; Behavioral: Education
- Education (Active Comparator): An activity diary and a pedometer will be given to write down the number of steps per day.
  After one week, the patient will be asked to send the activity diary as a photo via WhatsApp.
  Afterwards, a 20-minute phone call will be made to provide patient education.
  A reminder call will be made to the patient in the 4th week after the training and any questions will be answered.
  Individuals in the patient education group will be asked to record their steps for one week with a pedometer in the 8th week after the training.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Digitally assisted behavioral physical activity intervention — Digitally Assisted Behavioral Physical Activity Intervention Each week, the step count target will be renewed and an average of 20 minutes of phone calls will be made, including motivational interviews guided by Social Cognitive Theory. Motivational interviews will last 8 weeks.
  Outcome Expectations - Informing about the positive results when the physical activity level is increased and the dose-effect relationship Self Efficacy - Individuals' previous physical activity/exercise experiences will be evaluated and discussed.
  Social Support - A WhatsApp group will be created. Self Regulation - Self-monitoring ; Goal setting; Feedback, Self-reward
  Arms: Digitally assisted behavioral physical activity intervention+Education
Behavioral: Education — Patient Education
  * Definition of fibromyalgia syndrome
  * Symptoms of fibromyalgia syndrome
  * Exercise and physical activity
  * Recommendations to improve the quality of life
  * Sleep quality and sleep hygiene
  * Pain management
  * Fatigue and energy conservation techniques All patient education content will also be available on the website.

SUMMARY:
Digital health interventions have the potential to address physical inactivity as they are accessible to a large part of the population and can be delivered with high efficiency at a low cost. By enabling patient education, support for self-management, motivation, follow-up, feedback and communication, it can prevent, cure or treat many chronic conditions. These features can increase patient motivation and encourage compliance with home exercises and physical activity . Digital behavior change interventions use digital technologies (such as websites, mobile apps, Short Message Service or wearable devices) to promote and maintain health and have the potential to overcome many barriers compared to in-person programs by providing cost-effective, effective, and accessible information.

No study has been found in Turkey examining digital interventions or walking programs that include behavior change techniques to increase physical activity in patients with fibromyalgia syndrome. Considering environmental, cultural and economic factors in this patient group in our society, the investigators think that walking, which the investigators think is the most appropriate physical activity method in terms of cost, accessibility and equipment, should be a permanent behavior. The use of technology to increase physical activity in the era of digitalization is important in terms of addressing the increasing inactivity during the Covid19 pandemic period.

The aim of this study is to estimate the effect of digital assisted physical activity intervention combined with patient education compared to patient education alone on physical activity level, functional capacity, quality of life, sleep quality, pain, fatigue, and perspective on exercise of adults with Fibromyalgia Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having a female gender
* Reporting at least 40 mm in weekly pain intensity from the VAS scored between 0-100 with 'no pain' and 'worst possible pain'
* Using a fixed dose of medication for at least the past 6 months
* Being in the "Inactive" group according to the International Physical Activity Survey (not participating in physical activity to meet the physical activity recommendations of the guides)
* Using / agreeing to use WhatsApp application

Exclusion Criteria:

* Having another disease that affects the physical condition
* Cognitive inability to cooperate
* Being pregnant
* Inability to understand or speak Turkish
* Concurrent autoimmune or inflammatory disease,
* Diseases affecting the central nervous system (eg multiple sclerosis, Parkinson's disease),
* Serious psychiatric conditions that prevent participation (eg, psychotic disorders).
* Participation in a rehabilitation program in the past year,
* Exercising regularly for 6 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Step Counts at 2 months | At the baseline and 2 months later
  The pedometer is an inexpensive, easy-to-use instrument designed to measure the number of steps and walking distance, providing objective measurement. It is usually attached to the lumbar region and includes a lever arm connected to a horizontal spring that bounces off with the vertical acceleration of the hips during walking (up-down motion during cruising). Pedometers designed to detect vertical movement logically determine the number of steps. The output of the device is easily understood as the number of movements representing a step. The pedometer (pedometer) is an easy-to-use device that can be easily carried by people and can approximate the number of steps, the distance walked and the calories consumed.
Change from Baseline Physical Activity Level at 2 months | At the baseline and 2 months later
  The purpose of the questionnaire is to obtain data on health-related physical activity. We used the short self-administered version in the present study. The short form International Physical Activity Questionnaire (IPAQ) is a 9-item scale, assessing the amount of minutes spent in vigorous and moderate intense activity and walking during the last 7 days. Also the amount of minutes spending sitting on week days in the past 7 days is assessed. For all categories patients have to define on how many days and how many minutes they spent at a specific activity category. For all categories, the amount of Metabolic Equivalents (METs)-minutes is calculated by multiplying the amount of minutes with 8 (vigorous), 4 (moderate), 3.3 (walking), or 1.3 (sitting). Besides these four subscores, a total score is calculated by counting the METs-minutes of the first 3 categories together.

SECONDARY OUTCOMES:
Change from Baseline Functional Capacity at 2 months | At the baseline and 2 months later
  A chair without arms, with rubber tips on the legs, a hard seat of fixed height 46 cm was positioned against a wall. Test protocol required the participant to commence in a seated position with the feet resting flat and ankle joints in the neutral position. All participants were given the instruction to perform the sit-to-stand task as quickly as possible with their arms crossed over the chest and hands on the shoulders. A standard Sit to Stand (STS) movement was viewed as the legs being fully straightened when the stand phase concluded and the hip landing firmly on the chair when seated. A test would be terminated if the participant required assistance or was unable to complete the movement. No encouragement was provided during any STS test protocol.
  30 seconds STS tests, subjects were required to perform as many STS movements as possible within 30 seconds, respectively. The number of STS movements completed within the time required was recorded, as appropriate.
Change from Baseline Quality of Life at 2 months | At the baseline and 2 months later
  The Fibromyalgia Impact Questionnaire (FIQ) was developed in 1991, with subsequent modifications in 1997 and 2002. It has been validated as an effective tool for assessing status and function of patients with fibromyalgia.The FIQ is a self-administered instrument and contains ten questions that assess the following areas: physical functioning, symptoms of pain, fatigue, morning tiredness, stiffness, job difficulty, depression, anxiety, days of work missed, and overall well being in the previous week. The possible range of score is from 0 to 100, with a higher score indicating a greater effect of the syndrome on the individual.
Change from Baseline Sleep Quality at 2 months | At the baseline and 2 months later
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report measure of sleep quality over the previous month. It consists of seven component scores, each rated on a 0-3 scale, with higher scores implying greater difficulties. These seven component scores can be summed to form a single global score, which ranges from 0 to 21, with higher scores reflecting greater overall sleep disturbance. The PSQI has demonstrated adequate internal consistency, test-retest reliability, and discriminative validity in a mixed sample of participants ages 19-83 (M=49.5), with major depressive disorder, sleep disorders, or no psychiatric disorder. A global PSQI score of 5 or greater is indicative of poor sleep quality among younger adults, though others suggest a cut-off of 8.
Change from Baseline Pain at 2 months | At the baseline and 2 months later
  The visual analogical scale (VAS) is commonly employed to assess the perception of somatic pain intensity. Validated in fibromyalgia patients, this scale has a score from 0 to 10, where 0 refers to pain free or "no pain" and 10 refers to "worst possible pain". It is a single-item scale. Test-retest reliability has been shown to be good, but is higher among literate (R = 0.94, p < 0.001) than illiterate patients (R = 0.71, p < 0.001) before and after attending a rheumatology outpatient clinic.
Change from Baseline Fatigue at 2 months | At the baseline and 2 months later
  Fatigue severity scale (FSS); a Likert scale consisting of nine items that assess fatigue severity and functionality. Items were rated on a scale of 1 to 7 according to their level of agreement with a given statement and included statements such as "I am easily fatigued" or "Fatigue interferes with carrying out certain duties and responsibilities". Values for each item were averaged for a composite score, with higher scores indicating higher levels of impairment as a result of fatigue. FSS has been used in clinical practice for fatigue symptoms in people with chronic neck pain, showing high internal consistency (Cronbach's alpha > 0.8)
Change from Baseline Physical Activity Perception at 2 months | At the baseline and 2 months later
  Exercise Benefits/Barriers Scale (EBBS) is consisted of 42 items, 14 of the Barriers Scale and 28 of the Benefits Scale. This scale presents answer options of the Likert type with rating levels varying from one (1) to four (4): strongly agree (4), agree (3), disagree (2), strongly disagree (1). When used together, the EBBS has a reverse score of the items of the Barriers Scale, ranging from 42 until 168. Isolatedly, the highest score is of the Benefits Scales that ranges from 28 to 112 and of the Barriers Scale, from 14 until 56, representing the best perception of the benefits and the barriers respectively.
Change from Baseline Physical Activity Awareness at 2 months | At the baseline and 2 months later
  Physical activity awareness will be assessed with Cognitive Behavioral Physical Activity Questionnaire (CBPAQ). The CBPAQ scale consists of 15 items, including three sub-dimensions: personal barriers, outcome expectations and self-regulation. The individual items are rated at 1-5 according to the situation in which they are most appropriate. The higher the score, the higher the level of awareness.
Activity Diary | At the baseline and 2 months later
  The activity diary is a chart prepared in the form of weekly periods in which patients record their pedometer outputs (walking time, number of steps, walking distance) daily.

CONTACTS AND LOCATIONS:
Locations (1):
- Nimet Sermenli Aydın, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided